CLINICAL TRIAL: NCT01762202
Title: Phase 2 Multicenter, Study to Assess the Efficacy and the Safety of Front-line Fludarabine, Cyclophoshamide and Ofatumumab (FCO2) Chemoimmunotherapy in Young (≤65 Yrs) Patients With Chronic Lymphocytic Leukemia (CLL).
Brief Title: Assessment of Efficacy and Safety of Front-line Fludarabine, Cyclophoshamide and Ofatumumab Chemoimmunotherapy in Young Patients With Chronic Lymphocytic Leukemia.
Acronym: CLL0911
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL0911; 2011-005329-27 (EudraCT Number)
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: B-cell Lymphoid Leukemia; Young Patients
Keywords: CLL; Fludarabine; Cyclophosphamide; Ofatumumab
MeSH Terms: interventions — Cyclophosphamide; fludarabine; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study therapy (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Ofatumumab

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Fludarabine
Drug: Ofatumumab

SUMMARY:
Assessment of safety and efficacy of with fludarabine and cyclophosphamide (FC) combined with ofatumumab (FCO2) in previously untreated "young" patients with Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
Given that:

* rituximab, fludarabine and cyclophosphamide (FCR) front-line treatment was associated with a high OR rate, superior PFS and OS as compared to fludarabine and cyclophosphamide regimen;
* a direct relationship between the dose of rituximab and the response rate has been reported;
* ofatumumab, as single agent, proved activity in CLL patients with refractory disease;
* ofatumumab, fludarabine and cylophosphamide (O-FC) front-line treatment has been associated with a high complete response (CR) rate;
* the expected grade 3-4 granulocytopenia could led to reduce the dose intensity of study drugs (FC) and increase the infection rate; a schedule combining FC with an increased dose of ofatumumab associated to primary phrophylaxis of granulocytopenia could be associated with an improvement in the CR rate. The purpose of this study is to determine whether we could improve the CR rate of the golden standard treatment for fit patients with CLL , the FCR regimen, with a chemoimmunotherapy including FC combined with an increased dose of the monoclonal antibody ofatumumab, given every other week (FCO2) associated with a primary prophylaxis of granulocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* B-cell CLL diagnosis by 2008 revised IWCLL criteria.
* Treatment requirement according to the 2008 revised IWCLL criteria.
* No previous treatment.
* Age > 18 year and . 65 years.
* ECOG performance status of 0-1 at study entry and CIRS score .6.
* Adequate renal function (creatinine clearance.60 ml/min estimated using the Cockcroft-Gaultequation) .
* For male and female subjects of childbearing potential, agreement to use effective contraception.
* Signed written informed const according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease and/or laboratory abnormality which in the opinion of the investigator may represent a risk for the patient and/or that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Known positive serology for HIV.
* Positive serology for Hepatitis B (HBV) defined as a positive test for HBsAg and HBV-DNA.
* HCV-RNA positive.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection, tuberculosis and active hepatitis.
* History of tuberculosis within the last five years or recent exposure to tuberculosis equal to or less than 6 months.
* Known presence of alcohol and/or drug abuse.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to the inclusion in the study, congestive heart failure (NYHA III-IV), arrhythmia unless controlled by therapy.. grade 2 neuropathy; history of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* One or more laboratory abnormalities:

  1. Calculated creatinine clearance (Cockroft-Gault)<60mL/min.
  2. Absolute granulocyte count <1500/ƒÊL not disease related.
  3. Platelet count < 75000/ƒÊL not disease related.
  4. GOT, GPT, GT, alkaline phosphatase > 1,5 x upper limit of normal value unless due to disease involvement); serum bilirubin >1.5mg/dL, subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones)
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of complete responses. | After 8 months from study entry.
  The complete response (CR) rate after FCO2 front-line treatment.

SECONDARY OUTCOMES:
Number of overall responses. | After 8 months from study entry.
  Overall Response (OR) rate after FCO2 front-line treatment.
Number of patients in progression-free survival. | After 32 months from study entry.
  Progression-free survival (PFS) calculated from the date of first treatment dose - induction phase - until the date of the first documentation of progressive disease or until death (whatever the cause), whichever occurs first. Patients still alive and known to be progression free will be censored at the moment of last follow-up.
Number of patients needing a new CLL Treatment. | After 32 months from study entry.
  Time to a new CLL treatment (TTT) will be calculated from the date of last treatment dose until date of a new treatment received for CLL, where death occurred before the new treatment will be considered as competing risk. Patients still alive without receiving a new treatment will be censored at the time of the last follow-up.
Number of patients in overall survival | After 32 months from study entry.
  Overall survival (OS): defined as the time interval between the date of first treatment dose - induction phase- and the date of death for any cause; patients still alive will be censored at the moment of last follow-up.
Number of toxic events. | After 32 months from study entry.
  Toxicity of treatment according the last NCI criteria.
Outcome of patients according to clinical and biologica variables. | After 32 months from study entry.
  Outcome of patients (response, PFS OS) according to clinical and biologic variables (age; size of nodes, 2-microglobulin, lymphocyte count, stage, IgVH, p53, FISH, ZAP-70, CD38, FLCs).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Pr., Study Chair — Policlinico Umberto I, Hematology Department.; Francesca R. Mauro, Study Director — Policlinico Umberto I, Hematology Department.
Locations (22):
- Italy (22):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - S.O.C. di Medicina Interna B - Ospedale - Cardinal Massaia di Asti, Asti
  - ASL12 - Biella Ospedale degli Infermi - Dip. di Medicina e Geriatria - Struttura Complessa di Medicina Interna, Biella
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - RCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Ospedale Niguarda " Ca Granda", Milan
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Policlinico Umberto I, Hematology Department - Sapienza, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - SS.C. di Oncoematologia - Dipartimento di Medicina Clinica e Sperimentale - Azienda Ospedaliera - S. Maria Di Terni, Terni
  - Div. di Ematologia Ospedale "S.Giovanni Battista", Torino
  - Clinica Ematologica - Policlinico Universitario, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it